CLINICAL TRIAL: NCT04819490
Title: A UK Multicentre, Non-interventional, Observational, Health-Related Quality of Life Study for Children and Adolescents With X-linked Hypophosphataemia
Brief Title: A UK Multicentre, Health-Related Quality of Life Study for Children and Adolescents With XLH
Status: Completed | Type: Observational
Sponsor: Kyowa Kirin Pharmaceutical Development Ltd (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: 2020-55-UK-CRY
Record Dates: First submitted 2021-03-18; First posted 2021-03-29 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: X-Linked Hypophosphataemia
Keywords: Crysvita; Burosumab; X-linked Hypophosphataemia (XLH); PHEX Gene Mutation
MeSH Terms: conditions — Familial Hypophosphatemic Rickets

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to provide Health-related Quality of Life (HRQoL) data from children and adolescents with growing skeletons in the United Kingdom (UK), including those treated with burosumab or alternative XLH treatment, as part of an updated submission to the SMC in early 2023. This study will utilise data from a subset of UK sites already within the XLH Registry (including participating Scottish sites) and collect additional HRQoL data within these sites (that are otherwise not included in the wider XLH Registry protocol). The HRQoL data will enable the calculation of HRQoL to derive the HRQoL utility estimates in children and adolescents with growing skeletons for the RSS health states, hence addressing an area of uncertainty.

DETAILED DESCRIPTION:
This is a multicentre, non-interventional HRQoL study of children and adolescents with growing skeletons using routinely collected XLH Registry data and prospectively collected HRQoL data. This study will aim to enrol approximately 50 patients from approximately 5 UK centres (currently participating in the XLH Registry) over a 6-month period. Each patient will be followed for up to 12 months after enrolment. As stipulated, the data collection should not require additional patient visits or data collection within the health service.

Three types of data will be used in this study:

1. Routinely collected data from the XLH Registry on patient demographics and clinical data, as well as PedsQL HRQoL data.
2. HRQoL data prospectively collected at enrolment, 6-month and 12-month follow-up by the patient and/or their parent / legal guardian.
3. RSS scores within the XLH Registry will be used where available, or RSS will be centrally calculated retrospectively from radiographs of the affected wrist and/or knee. All RSS calculations will be centrally reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥4 years and <18 years.
2. Enrolled in the XLH Registry via one of the participating UK centres.
3. Have at least one of the following:

   1. RSS calculated at enrolment during a routine clinic visit. OR
   2. Historical radiographs of the affected wrist and/or knee available in the medical chart within the 6 months prior to enrolment, to allow RSS to be centrally calculated retrospectively.
4. Receiving any XLH treatment (burosumab, oral phosphate and active vitamin D, or other XLH treatment) within 30 days prior to informed consent for this study

Exclusion Criteria:

1. Does not have the cognitive capacity to provide informed consent, or their legally designated representative (i.e. parent / legal guardian) does not have the cognitive capacity to provide informed consent.
2. Is not expected to have open growth plates for the duration of the study.
3. Currently participating in an interventional clinical trial. Participation in a Compassionate Use Programme, Pre-commercial Programme, or Investigator Initiated Study does not preclude a patient from participation in this study.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will aim to enrol approximately 50 patients from at least 5 UK centres (currently participating in the XLH Registry).
  Subjects will be receiving any XLH treatment (burosumab, oral phosphate and active vitamin D or another XLH treatment) within 30 days or prior to informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
To derive health state utilities based on Rickets Severity Score (RSS), in the study population | Changes from baseline, 6 months and 12 months
  The RSS is a quantitative method to assess rickets severity in the wrists and knees based on the degree of metaphyseal fraying, concavity, and the proportion of the growth plate affected. It is a 10-point scale, where 10 represents the most extreme degree of rickets severity. In nutritional rickets, RSS may range from 0.5 to 10.
To derive health state utilities based on EQ-5D-Y in the study population | Changes from baseline, 6 months and 12 months
  The EQ-5D-Y is a two-part instrument: the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system covers five health domains: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each domain has 3 response categories: no problems, some problems and a lot of problems. The response categories can be reflected by a 1-digit number (1-3) and combined for the five dimensions into a 5-digit number to describe the health state of the patient. The EQ VAS records the patient's self-rated health on a vertical VAS of 0-100 where 100="The best health you can imagine" and 0="The worst health you can imagine". The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement; results can be presented as both a measure of the central tendency and a measure of dispersion.
To derive health state utilities based on Child Health Utility 9 Dimensions [CHU-9D], in the study population | Changes from baseline, 6 months and 12 months
  CHU-9D is a generic child HRQoL questionnaire consisting of nine items, each with five response categories. Each item covers a different domain: worry, sadness, pain, tiredness, annoyance, school, sleep, daily routine and activities.

CONTACTS AND LOCATIONS:
Overall Officials: Kyowa Kirin Medical Affairs Division, Study Director — Kyowa Kirin, Inc.
Locations (6):
- United Kingdom (6):
  - Royal Hospital for Sick Children, Edinburgh
  - NHS Greater Glasgow & Clyde- South Glasgow University Hosp Division, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Trust Headquarters, St. James's University Hospital, Leeds
  - Evelina Childrens Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Sheffield Childrens Hospital, Sheffield